CLINICAL TRIAL: NCT02655081
Title: Investigating the Use of a Preoperative High-Arginine Nutritional Supplement Prior to Radical Cystectomy
Acronym: IMPACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Tatum Tarin, MD, Clinical Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO13060027
Record Dates: First submitted 2015-12-09; First posted 2016-01-13 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Bladder Cancer
Keywords: Urinary diversion; Bladder Neoplasm; Nutritional Supplement; Cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary supplement (Experimental): Subjects will receive high arginine nutritional supplement (Nestle's Impact AR), prior to cystectomy
  Interventions: Dietary Supplement: high arginine nutritional supplement (Nestle's Impact AR)

INTERVENTIONS:
Dietary Supplement: high arginine nutritional supplement (Nestle's Impact AR) — Preoperative High-Arginine Nutritional Supplement Prior to Radical Cystectomy

SUMMARY:
To provide patients with bladder cancer who are scheduled to undergo radical cystectomy with a preoperative high-arginine nutritional supplement. The investigator will measure patient adherence to the regimen, tolerability of the supplement and feasibility of supplementation. Secondary outcome measures will include differences in length of stay and complication rate between groups.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the use of a high-arginine protein supplement prior to surgery for patients undergoing radical cystectomy for treatment of bladder cancer. As many as 50% of patients who undergo radical cystectomy experience a postoperative complication, and poor preoperative nutritional status is known to increase the risk of complications. Preoperative use of a high-arginine protein shake has been shown to reduce the risk of postoperative complications for patients undergoing surgery for colon cancer, and this study seeks to determine whether this is also true for patients undergoing radical cystectomy for bladder cancer.

Subjects will drink four protein shakes (Nestle Impact AR) per day for 5-7 days prior to radical cystectomy. Shakes will be provided to patients free of charge. On the date of surgery, subjects will turn in a log of shake consumption. Surgery will then proceed in typical fashion, and no changes will be made to surgery or postoperative care. Clinical outcomes for the first 90 postoperative days will be collected. Patient outcomes will be compared to those of contemporary controls who do not undergo supervised nutritional supplementation. Primary study outcome is to assess safety, tolerability and adherence to supplementation regimen. Secondary outcomes include differences in complication rates and length of postoperative hospital stay between groups.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient seen at one of the aforementioned UPMC facilities who carries a diagnosis of bladder cancer and is considered a candidate for radical cystectomy for treatment.

Exclusion Criteria:

* Minors < 18 years of age, patients not considered surgical candidates, patients who do not go on to undergo radical cystectomy. Patients with Glomerular Filtration Rate (GFR) < 30 will also be excluded in an attempt to limit protein intake of patients with Stage IV and V Chronic Kidney Disease. Diabetic patients will be allowed to participate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and adherence to supplementation regimen." | 4 months
  Investigator will report on any adverse events from supplementation as well as patient adherence to regimen.

SECONDARY OUTCOMES:
Incidence of 90-day overall and infectious complication rates. I | 4 months
  Investigator will compare overall, infectious and wound complication rates between the study group and control group
Length of hospital stay between study group and control group | 4 months
  The Investigator will compare the length of hospital stay between study group and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Tatum Tarin, MD, Principal Investigator — Associate Professor of Medicine
Locations (1):
- Shadyside Urology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Braga M, Gianotti L, Radaelli G, Vignali A, Mari G, Gentilini O, Di Carlo V. Perioperative immunonutrition in patients undergoing cancer surgery: results of a randomized double-blind phase 3 trial. Arch Surg. 1999 Apr;134(4):428-33. doi: 10.1001/archsurg.134.4.428. PMID 10199318
- [Background] Shabsigh A, Korets R, Vora KC, Brooks CM, Cronin AM, Savage C, Raj G, Bochner BH, Dalbagni G, Herr HW, Donat SM. Defining early morbidity of radical cystectomy for patients with bladder cancer using a standardized reporting methodology. Eur Urol. 2009 Jan;55(1):164-74. doi: 10.1016/j.eururo.2008.07.031. Epub 2008 Jul 18. PMID 18675501
- [Background] Lee CT, Madii R, Daignault S, Dunn RL, Zhang Y, Montie JE, Wood DP Jr. Cystectomy delay more than 3 months from initial bladder cancer diagnosis results in decreased disease specific and overall survival. J Urol. 2006 Apr;175(4):1262-7; discussion 1267. doi: 10.1016/S0022-5347(05)00644-0. PMID 16515975
- [Background] Gibbs J, Cull W, Henderson W, Daley J, Hur K, Khuri SF. Preoperative serum albumin level as a predictor of operative mortality and morbidity: results from the National VA Surgical Risk Study. Arch Surg. 1999 Jan;134(1):36-42. doi: 10.1001/archsurg.134.1.36. PMID 9927128
- [Background] Gregg JR, Cookson MS, Phillips S, Salem S, Chang SS, Clark PE, Davis R, Stimson CJ Jr, Aghazadeh M, Smith JA Jr, Barocas DA. Effect of preoperative nutritional deficiency on mortality after radical cystectomy for bladder cancer. J Urol. 2011 Jan;185(1):90-6. doi: 10.1016/j.juro.2010.09.021. Epub 2010 Nov 12. PMID 21074802
- [Background] Hollenbeck BK, Miller DC, Taub DA, Dunn RL, Khuri SF, Henderson WG, Montie JE, Underwood W 3rd, Wei JT. The effects of adjusting for case mix on mortality and length of stay following radical cystectomy. J Urol. 2006 Oct;176(4 Pt 1):1363-8. doi: 10.1016/j.juro.2006.06.015. PMID 16952633
- [Background] Waitzberg DL, Saito H, Plank LD, Jamieson GG, Jagannath P, Hwang TL, Mijares JM, Bihari D. Postsurgical infections are reduced with specialized nutrition support. World J Surg. 2006 Aug;30(8):1592-604. doi: 10.1007/s00268-005-0657-x. PMID 16794908
- [Background] Braga M, Gianotti L, Vignali A, Carlo VD. Preoperative oral arginine and n-3 fatty acid supplementation improves the immunometabolic host response and outcome after colorectal resection for cancer. Surgery. 2002 Nov;132(5):805-14. doi: 10.1067/msy.2002.128350. PMID 12464864
- [Background] Schiesser M, Kirchhoff P, Muller MK, Schafer M, Clavien PA. The correlation of nutrition risk index, nutrition risk score, and bioimpedance analysis with postoperative complications in patients undergoing gastrointestinal surgery. Surgery. 2009 May;145(5):519-26. doi: 10.1016/j.surg.2009.02.001. Epub 2009 Mar 27. PMID 19375611
- [Background] Oh CA, Kim DH, Oh SJ, Choi MG, Noh JH, Sohn TS, Bae JM, Kim S. Nutritional risk index as a predictor of postoperative wound complications after gastrectomy. World J Gastroenterol. 2012 Feb 21;18(7):673-8. doi: 10.3748/wjg.v18.i7.673. PMID 22363139
- [Background] Giger U, Buchler M, Farhadi J, Berger D, Husler J, Schneider H, Krahenbuhl S, Krahenbuhl L. Preoperative immunonutrition suppresses perioperative inflammatory response in patients with major abdominal surgery-a randomized controlled pilot study. Ann Surg Oncol. 2007 Oct;14(10):2798-806. doi: 10.1245/s10434-007-9407-7. Epub 2007 Jul 15. PMID 17632760